CLINICAL TRIAL: NCT02914977
Title: A Pilot Study of Low-Dose Daunorubicin in Patients With Relapsed/Refractory Acute Leukemia
Brief Title: Low-Dose Daunorubicin in Relapsed/Refractory Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tara Lin (Other)
Responsible Party: Sponsor-Investigator, Tara Lin, Medical Doctor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2016-RP-HEM-LD-DNR
Record Dates: First submitted 2016-07-25; First posted 2016-09-26 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Acute Lymphocytic Leukemia; Acute Myeloid Leukemia
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Recurrence | interventions — Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low-dose daunorubicin (DNR) (Experimental): Eligible patients will be treated with 5 days of low dose daunorubicin (DNR) for one cycle only.
  Interventions: Drug: Daunorubicin

INTERVENTIONS:
Drug: Daunorubicin — * Agent: Daunorubicin
  * Dose: 6.75 mg/m2/day
  * Route: IV
  * Schedule: Days 1-5
  * Duration: One cycle
  Other Names: Cerubidine; Daunoxome

SUMMARY:
In this pilot study, eligible patients will be treated with 5 days of low dose daunorubicin for one cycle only. Any patient who receives treatment on this protocol will be evaluable for toxicity. Each patient will be assessed for the development of toxicity at all scheduled visits (Days 1-5). Following participation on this brief pharmacodynamic trial, patients can then proceed to other conventional or investigational therapies, as clinically indicated.

DETAILED DESCRIPTION:
Disease relapse remains the primary challenge in the treatment of acute myeloid leukemia (AML) and acute lymphocytic leukemia (ALL). There is no standard of care treatment option for relapsed acute leukemia, and investigational therapies are recommended. Clinically targeting the leukemia stem cell (LSC) remains an unmet need in both AML and ALL. Therefore, a primary objective of this trial is to determine the molecular pharmacodynamic effects of low dose daunorubicin (DNR) on beta-catenin phosphorylation in serial bone marrow samples of patients with relapsed leukemia.

Prior to studying low-dose DNR in complex, multi-agent regimens, it is essential to confirm that it inhibits p-beta-catenin S552 in humans. This pilot study is designed to assess the feasibility and tolerability of low dose DNR administration to patients with relapsed/refractory AML and ALL, and obtain preliminary data regarding target engagement. A second objective is to demonstrate the safety and feasibility of low-dose daunorubicin administration in patients with relapsed/refractory acute leukemia.

Beta-catenin phosphorylation will be measured by immunohistochemistry assay in bone marrow samples taken from patients at study entry and at Day 8 following study therapy with low-dose DNR. The investigators will also measure the pharmacokinetics of low dose DNR in these patients, to enable preliminary PK-PD analyses and because there are essentially no PK data for DNR at comparable doses using modern analytical methodologies.

Following participation on this brief pharmacodynamic proof-of-concept trial, patients can then proceed to other conventional or investigational therapies, as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent or have parental consent.
* Age ≥ 18 years
* Pathological confirmation by bone marrow documenting the following:

  1. AML which has relapsed after Complete Remission
  2. AML which has been refractory to two prior induction attempts
  3. ALL which has relapsed after Complete Remission
  4. ALL which has been refractory to two prior induction attempts
* Disease status allows delay of additional anti-leukemia therapy for the duration of the study (hydroxyurea is allowed for control of WBC throughout study)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-3
* Able to adhere to the study visit schedule and other protocol requirements
* Cardiac ejection fraction ≥45% by ECHO
* Serum alanine aminotransferase or aspartate aminotransferase < 3 times the ULN
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

Exclusion Criteria:

* Concurrent use of conventional or investigational anticancer agents, except hydroxyurea (Standard prophylactic anti-infectives and medications to prevent/treat tumor lysis syndrome are allowed. Hydroxyurea may be used to keep the WBC<25,000. Additional anti-leukemia therapy is prohibited during the study.).
* Patient has received chemotherapy or radiotherapy within 2 weeks prior to entering the study or has not recovered from adverse events due to agents administered more than 2 weeks earlier, with the exception of hydroxyurea.
* Patients with known active uncontrolled central nervous system (CNS) leukemia
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to daunorubicin
* Patients with a total lifetime anthracycline exposure exceeding the equivalent of 900 mg/m2 of daunorubicin
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Unwilling or unable to undergo serial bone marrow aspirate/biopsy
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Molecular pharmacodynamic effect of low dose daunorubicin on beta-catenin phosphorylation as assessed by quantitative immunohistochemistry assay performed on serial bone marrow samples of patients with relapsed leukemia. | 12 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events and/or toxicity as assessed by CTCAE 4.03. | 12 months
  Analyses will be performed for all patients having received at least one dose of study drug. Each patient will be assessed for the development of toxicity at all scheduled visits (Days 1-5).
Maximum Plasma Concentration [Cmax] | prior to dosing and 5, 20, and 40 min and 1, 2, 4, 8, and 24 hrs after dosing
Area Under the Curve [AUC] | prior to dosing and 5, 20, and 40 min and 1, 2, 4, 8, and 24 hrs after dosing

OTHER OUTCOMES:
Test for additional validated markers for leukemia and/or stem cells (such as anti-CD34 and CD38, CD45 and/or CD19) assessed by flow cytometry of serial bone marrow samples. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tara Lin, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Cancer Center - Clinical Research Center, Fairway, Kansas, United States